CLINICAL TRIAL: NCT05989334
Title: Kayseri City Hospital
Brief Title: Epidemiological Data of Patients Consulted to Kayseri City Hospital Physical Therapy Clinic in the 2023 Kahramanmaraş Earthquake
Status: Completed | Type: Observational
Sponsor: Kayseri Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Ayşe Güç, physical medicine and rehabilitation, Kayseri Education and Research Hospital
Other Study IDs: 0000-0003-2552-1403
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: in the Writing Process
Keywords: 2023 Kahramanmaraş, earthquake

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The quality of life of people after the earthquake is significantly affected. In particular, adequate and correct management of the damage caused by trauma on the human body is very important to reduce disability. Epidemiological information about the injury pattern from past earthquakes is crucial for preparedness and effective response to potential earthquakes in regions where resources are scarce. Thanks to the epidemiological data obtained from post-earthquake injury patterns, hospitals can be prepared for possible earthquakes, and disability and mortality can be reduced.

Although many earthquake victims suffer injuries that require treatment, there are large gaps in knowledge regarding the epidemiology of earthquakes. It is essential to evaluate the data collected after the earthquake in the planning phase of the health demands of the earthquake area. Epidemiological studies on earthquakes guide the planning and organization of health services for hospitals located in and around the earthquake area. By knowing the injury patterns that will occur after the earthquake, the effectiveness of the early and specific treatments to be applied to the earthquake victims can be increased significantly. In this way, complications, disability and mortality rates that may occur in future natural disasters can be reduced. The aim of this study is to record the injury patterns and treatments of the patients who were consulted to the physical therapy and rehabilitation clinic after the 2023 Kahramanmaraş earthquake in our country, which is an earthquake zone, and to ensure that the physical therapy physicians meet the possible earthquakes in a more knowledgeable, experienced and prepared manner.

ELIGIBILITY:
Inclusion Criteria:

* All age group patients, male and female, who had earthquake-related injuries and were consulted to the physical therapy unit were included in our study. Our study included both earthquake survivors who were consulted before the study (their files were scanned retrospectively) and newly registered patients (by obtaining voluntary consent form signatures).

Exclusion Criteria:

-

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 220 patients who were hospitalized due to injury and illness due to the 2023 Kahramanmaraş earthquake and were consulted to the physical therapy unit were examined.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Epidemiological Data of Patients Consulted to Kayseri City Hospital Physical Therapy Clinic in the 2023 Kahramanmaraş earthquake | 2023 February-2023 June

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri City Hospital, Kayseri, Turkey (Türkiye)